CLINICAL TRIAL: NCT01167231
Title: Acarbose in Cardiovascular Risk Management. Assessment of Clinical Efficacy and Safety of Acarbose and Its Effect on Selected Cardiovascular Risk Factors in Type 2 Diabetes Patients.
Brief Title: Prevention of Postprandial Hyperglycemia by Acarbose May be a Promising Therapeutic Strategy for Reducing the Increased Risk for Cardiovascular Disease
Acronym: ABDOMEN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Sp. z o.o.
Other Study IDs: 13066; GB0710PL
Record Dates: First submitted 2010-07-16; First posted 2010-07-22 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Acarbose
MeSH Terms: conditions — Diabetes Mellitus | interventions — Acarbose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)

INTERVENTIONS:
Drug: Acarbose (Glucobay, BAYG5421) — Patients treated with acarbose tablets under the real-life setting. Dosing regimen customised to the needs of each participating patient according to the investigators assessment

SUMMARY:
The use of acarbose in impaired glucose tolerance (IGT) and type 2 diabetic subjects has been associated with a significant reduction of cardiovascular events. Additionally, acarbose has been shown to have a beneficial influence on some of the other cardiovascular risk factors (metabolic syndrome components). Thus, prevention of postprandial hyperglycemia by acarbose may be a promising therapeutic strategy for reducing the increased risk for cardiovascular disease. Further studies are needed to confirm the influence of acarbose on cardiovascular risk factors in the real life setting.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus
* Age >/= 18 years
* Naive to acarbose (minimum 3 months before inclusion)

Exclusion Criteria:

* Hypersensitivity to acarbose or any of the excipients
* Age <18 years
* Pregnancy and in nursing
* Inflammatory bowel disease, colonic ulceration, partial intestinal obstruction or in patients predisposed to intestinal obstruction
* Chronic intestinal diseases associated with marked disorders of digestion or absorption
* States which may deteriorate as a result of increased gas formation in the intestine, (e.g. Roemheld's syndrome [an angina pectoris-like syndrome or aggravation of an angina pectoris due to the postprandial filling of the stomach] and larger hernias)
* Hepatic and severe renal impairment (creatinine clearance <25 mL/min/ 1,73m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic diabetic patients not treated with acarbose for at least 3 months.
Sampling Method: Probability Sample
Enrollment: 3310 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability of acarbose and its effect on body weight, waist circumference and blood pressure | approximately 6 months after acarbose treatment initiation

SECONDARY OUTCOMES:
Effect of acarbose on HbA1c, fasting and postprandial glycemia and on lipid profile | approximately 6 months after acarbose treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland